CLINICAL TRIAL: NCT01295411
Title: Morphological, Structural and Functional Neural Substrates of Quality of Life in Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A01421-38; 2010-29 (Other: AP HM)
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- schizophrenia PATIENTS (Other)
  Interventions: Device: Magnetic Resonance Imaging; Other: EVALUATION NEUROPSYCHOLOGICAL

INTERVENTIONS:
Device: Magnetic Resonance Imaging
Other: EVALUATION NEUROPSYCHOLOGICAL

SUMMARY:
The aim of the investigators analysis is to identify the neural correlates of quality of life scores in schizophrenia. For this, the investigators will constitute group of patients according to their quality of life scores and the investigators will analyze their differences in patterns of brain structures and activations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria (American Psychiatric Association(APA), 1994),
* age over 18 years,
* informed consent to participate in the studies
* French as native language

Exclusion Criteria:

* diagnosis other than schizophrenia on Axis I of DSM-IV,
* decompensated organic disease and mental retardation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
to study the relationships between quality of life and the morphologic, structural and functional substrates in schizophrenia | 36 months

SECONDARY OUTCOMES:
to determine whether quality of life is correlated with brain modifications using functional Magnetic Resonance Imaging | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Faget-Agius C, Boyer L, Wirsich J, Ranjeva JP, Richieri R, Soulier E, Confort-Gouny S, Auquier P, Guye M, Lancon C. Neural substrate of quality of life in patients with schizophrenia: a magnetisation transfer imaging study. Sci Rep. 2015 Dec 3;5:17650. doi: 10.1038/srep17650. PMID 26632639